CLINICAL TRIAL: NCT03433859
Title: Prospective Multicentric Open Randomised Controlled Trial Comparing Topical Aluminium Chloride to OnabotulinumtoxinA Intradermal Injections in Residual Limb Hyperhidrosis (Lower Limbs)
Brief Title: Topical Aluminium Chloride vs OnabotulinumtoxinA Intradermal Injections in Residual Limb Hyperhidrosis (Lower Limbs)
Acronym: SALUTOX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013RC09; 2014-002068-34 (EudraCT Number)
Record Dates: First submitted 2016-10-19; First posted 2018-02-15 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Hyperhidrosis; Residual Limbs
MeSH Terms: conditions — Hyperhidrosis | interventions — Botulinum Toxins, Type A; Aluminum Chloride; Cosmetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OnabotulinumtoxinA (Experimental): OnabotulinumtoxinA in intradermal Injections on residual lower limb
  Interventions: Drug: OnabotulinumtoxinA
- Topical Aluminium Chloride (Active Comparator): Topical Aluminium Chloride (cosmetic product) on the lower limb
  Interventions: Other: Topical Aluminium Chloride (cosmetic product)

INTERVENTIONS:
Drug: OnabotulinumtoxinA — OnabotulinumtoxinA in intradermal Injections on residual lower limb : 100 Units - 1 dose
  Other Names: Botox
  Arms: OnabotulinumtoxinA
Other: Topical Aluminium Chloride (cosmetic product) — Topical Aluminium Chloride (cosmetic product) : 1 quantity sufficient on the lower limb
  Arms: Topical Aluminium Chloride

SUMMARY:
The aim of this study is to demonstrate onabotulinumtoxinA superiority to aluminium chloride for the treatment of residual limb hyperhidrosis.

DETAILED DESCRIPTION:
After randomization patients will receive either OnabotulinumtoxinA once or topical aluminium chloride for 6 months. All patients will be evaluated during 3 study visits (week 4, week 12, week 24) and 1 phone call (week 18).

ELIGIBILITY:
Inclusion Criteria:

* Lower limb amputees suffering from residual limb hyperhidrosis with important cutaneous, functional, social and professional consequences, whatever the amputation cause
* HDSS ≥ 2 (Hyperhidrosis Disease Severity Score)
* Men and women
* 18 to 75 years old
* Written informed consent
* No exclusion criteria
* Social assurance

Exclusion Criteria:

* Botulinum toxin injection necessity for another disease
* Evolutive Central neurologic disease or myasthenia.
* Egg or albumine allergy
* Botulinum toxin or other excipients hypersensibility
* Legally protected Adults and people unable to give an informed consent. (article L-1121-8 from Public Health Code), people without freedom and people hospitalized without consent (article L-1121-6 from Public Health Code)
* Pregnant women or giving breast women (article L-1121-5 from Public Health)
* Patient refusing participating
* Previous hyperhidrosis treatment with aluminium chloride in the last 4 weeks
* Previous hyperhidrosis treatment with botulinum toxin in the last 2 years
* Other ongoing hyperhidrosis treatment
* Large residual limb eczematiform lesions: corticoids treatment (for example: Locapred® 1 application per day during 1 week then decrease).
* Aminoglycoside ongoing treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-03; Primary Completion 2020-09-10 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Hyperhidrosis Disease Severity Score (HDSS) evolution | 24 weeks
  HDSS score : min 1 - max. 4
  * Efficacy : HDSS evolution from 2 (initial measure) to 1 (final measure), from 3 (initial measure) to 1 or 2 (final measure), from 4 (initial measure) to 1 or 2 (final measure)
  * Failure : from 2 (initial measure) to 2 (final measure), from 3 or 4 (initial measure) to 2 (final measure) ; or increase of HDSS between initial and final measure

SECONDARY OUTCOMES:
Mismatch of prothesis associated with sweat measured by a visual analogue scale | 3 years
  Visual analogue scale (VAS) using 100mm scale. VAS range from 0 to 100mm. Efficacy is considered if > 50% increase between initial and final measure
Problems with walking due to sweat measured by a visual analogue scale | 3 years
  Visual analogue scale (VAS) using 100mm scale. VAS range from 0 to 100mm. Efficacy is considered if > 50% increase between initial and final measure
Sweat quantity measured by a visual analogue scale | 3 years
  Visual analogue scale (VAS) using 100mm scale. VAS range from 0 to 100mm. Efficacy is considered if > 50% increase between initial and final measure
Quality of life measured by a visual analogue scale | 3 years
  Visual analogue scale (VAS) using 100mm scale. VAS range from 0 to 100mm. Efficacy is considered if > 50% increase between initial and final measure
Amount of time spent wearing the prothesis | 3 years
  Amount of time spent wearing the prosthesis (hours per day): efficacy if increase
Prothesis removed to dry the residual limb | 3 years
  Number of times the prosthesis had to be removed to dry the residual limb and sleeve per day: efficacy if no need to remove it or only once a day
Quality of life(DLQI) | 3 years
  DLQI quality of life questionnaire : efficacy if increase
Quality of life (physical domain of SF36) | 3 years
  SF36 "limitations due to physical state" specific domain : efficacy if increase
Quality of life (subjective improvement felt) | 3 years
  Subjective Improvement Felt (SIF) (based on a percentage scale) :efficacy if>50% increase

CONTACTS AND LOCATIONS:
Overall Officials: Hélène BISSERIEX, MD, Principal Investigator — Service de Santé des Armées, Hôpital Clermont-Tonnerre (Brest, France)
Locations (9):
- France (9):
  - Les Capucins, Angers
  - Hôpital Clermont-Tonnerre, Brest
  - CMPR La Tour de Gassies, Bruges
  - Hopital Percy, Clamart
  - Hopital Laveran, Marseille
  - Pôle Saint Helier, Rennes
  - Centre La Tourmaline, Saint-Herblain
  - Institut Universitaire de Réadaptation Clémenceau, Strasbourg
  - Institut Robert Merle d'Aubigné, IRMA, Valenton

IPD SHARING:
Plan to Share IPD: No